CLINICAL TRIAL: NCT04234438
Title: Management of Cystoid Macular Edema Secondary to Retinitis Pigmentosa Via Subliminal Micropulse Yellow Laser
Acronym: SL-MPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principle investigator, MD, Ankara Universitesi Teknokent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1249-17
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Retinitis Pigmentosa; Cystoid Macular Edema
Keywords: Retinitis pigmentosa; Cystoid macular edema; Intraretinal cysts; Subliminal micropulse laser
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Edema

STUDY DESIGN:
Intervention Model Description: Prospective open-label clinical trial, included 32 eyes of 29 patients who had cystoid macular edema secondary to retinitis pigmentosa. Patients were treated by subliminal micropulse yellow laser for one session. Central macular thickness and best corrected visual acuity changes were investigated just before the treatment and 1 year later after the one session of the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Before application (Active Comparator): 32 eyes of 29 patients who had cystoid macular edema secondary to retinitis pigmentosa Before subliminal micropulse laser application
  Interventions: Device: SL-MPL treatment protocol was performed with a 577 nm yellow laser (EasyRet, Quantel Medical, Cedex, France)
- After application (Active Comparator): 32 eyes of 29 patients who had cystoid macular edema secondary to retinitis pigmentosa After 12 months subliminal micropulse laser application
  Interventions: Device: SL-MPL treatment protocol was performed with a 577 nm yellow laser (EasyRet, Quantel Medical, Cedex, France)

INTERVENTIONS:
Device: SL-MPL treatment protocol was performed with a 577 nm yellow laser (EasyRet, Quantel Medical, Cedex, France) — Macular laser treatment was applied after pupil dilation and topical anesthesia. Laser application was performed with a Mainster Standard contact laser lens (Volk Optical, Mentor, OH, USA). To determine the appropriate personalized calibration value, single-spot test shot was applied under the green filter to a non-edematous area of the macula outside the temporal vascular arcade. The laser power was gradually increased until it formed a barely visible laser spot. The power of the micropulse pattern laser was set at 50% of the power needed to form a barely visible laser spot. Laser parameters used were 200 ms duration, 160 µm spot diameter, low operating cycle (5%), and zero spacing with 5x5 pattern shape. SL-MPL was applied to the areas where edema was detected in OCT and examination.

SUMMARY:
Purpose: To investigate the effects of subliminal micropulse yellow laser application on central macular thickness and best corrected visual acuity in cystoid macular edema secondary to retinitis pigmentosa patients.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a progressive photoreceptor and retinal pigment epithelial (RPE) degeneration that begins as a night vision loss, resulting in narrowing of the visual field and legal blindness. RP is a heterogeneous genetic disorder, affecting 1/3000- 8000 people worldwide. RP is the result of mutation in one of more than 260 genes. These genes are responsible for the synthesis of peptides involved in the visual cycle. These genes are also responsible for the synthesis of growth factors responsible for the conversion of glucose to adenosine triphosphate (ATP) or responsible for the removal of metabolic wastes.

The incidence of cystoid macular edema (CME) in RP has been reported as between 10% - 50%. There are several hypotheses about the pathogenesis of cystoid macular edema in RP. The first hypothesis is explained by Müller cell hypertrophy and its paracrine effects. Mutations in the retinal pigment epithelium disrupt the synthesis of some growth factors. Stress caused by apoptosis in rod cells in the periphery leads to ectopic synaptogenesis of Müller cells in the central. Müller cells undergo copensatory hypertrophy and synthesize excessive growth factors. This paracrine effect provides protection of central vision. Edema in a certain level is considered to be protective to photoreceptors and should not be treated. But if edema is excessive and prolonged leads to a break in synaptic connections in the neural retina and an increase in neurodegeneration. CME also deteriorates central visual quality in patients with impaired peripheral vision. Treatment should be considered only if the edema is excessive and disrupts central vision. According to our clinical experience, when central macular thickness exceeds 500 microns, central visual quality of the patient decreases and requires treatment.

Other pathophysiological causes of CME in RP are explained by low grade inflammation and retinal autoantibodies. In some genetic mutation types of RP, such as the X-linked RPGR gene mutation; vitritis, lipofuscin deposits and inflammation are predominant. Ciliopathy leads to inflammation and CME, which increases photoreceptor loss rate. Immediate treatment of inflammation-induced edema can slow disease progression. Inflammatory edema appears as cystoid macular edema, whereas compensatory edema due to Müller cell hypertrophy is seen as separeted intraretinal cysts. Inflammatory edema responds well to carbonic anhydrase inhibitors, while compensatory edema does not.

The results of the treatment of CME in RP are controversial, as the compensatory or inflammatory distinction is not made clearly. Treatments such as grid laser photocoagulation, oral acetazolamide, topical carbonic anhydrase inhibitors, intravitreal therapy with corticosteroids or anti-vascular endothelial growth factor agents and pars plana vitrectomy may be effective in some cases with CME secondary to RP. Most of these treatments have either insufficient response or excessive side effects.

To our knowledge, so far, we have not found a scientific publication about the use of micropulse yellow laser for treatment cystoid macular edema secondary to retinitis pigmentosa.

Subliminal micropulse laser (SL-MPL) is a method developed to reduce the laser-induced thermal damage caused by conventional laser therapy for treatment some macular diseases. In the micropulse mode, laser is applied in short pulses, thereby reducing the thermal energy generated in the target area. The coagulation scars do not form with SL-MPL treatment. Sublethally injured RPE cells induce an up- and down regulation of various growth factors (GFs) [pigment epithelium-derived factor (PEDF), vascular endothelial growth factor (VEGF) inhibitors, VEGF inducers, permeability factors, etc.] which restores the pathologic imbalance.

The aim of this study was to investigate the effect of yellow (577 nm) SL-MPL therapy on central macular thickness (CMT) and on best corrected visual acuity (BCVA) in patients with cystoid macular edema secondary to retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any phenotypic variation of RP
* Presence of separeted intraretinal cysts
* Central macular thickness ≥ 500 µm
* Unresponsive to systemic or topical carbonic anhydrase inhibitors
* No interventional treatment for macular edema in the last 3 months

Exclusion Criteria:

* Patients with signs of inflammation, such as cells in the vitreous, intraretinal white dots, septa-free edema
* Patients responding to systemic or topical carbonic anhydrase inhibitors
* Any interventional treatment has been applied for macular edema in the last 3 months
* The presence of other causes that may lead to CME such as epiretinal membrane, vitreous traction, diabetes or uveitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | Change from baseline central macular thickness at 12 months
  It is obtained by measuring the distance between the internal limiting membrane and the bruch membrane in the center of fovea by OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Arslan, MD, Principal Investigator — Ankara Universitesi Teknokent
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University Biotechnology Institute, Ankara, Türkiye
  - Umut Arslan, Ankara, Türkiye

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakthavatchalam M, Lai FHP, Rong SS, Ng DS, Brelen ME. Treatment of cystoid macular edema secondary to retinitis pigmentosa: a systematic review. Surv Ophthalmol. 2018 May-Jun;63(3):329-339. doi: 10.1016/j.survophthal.2017.09.009. Epub 2017 Oct 5. PMID 28987613
- [Result] Scholz P, Altay L, Fauser S. A Review of Subthreshold Micropulse Laser for Treatment of Macular Disorders. Adv Ther. 2017 Jul;34(7):1528-1555. doi: 10.1007/s12325-017-0559-y. Epub 2017 May 24. PMID 28540655
- [Result] Luttrull JK. Improved retinal and visual function following panmacular subthreshold diode micropulse laser for retinitis pigmentosa. Eye (Lond). 2018 Jun;32(6):1099-1110. doi: 10.1038/s41433-018-0017-3. Epub 2018 Feb 16. PMID 29449615
- [Derived] Arslan U. Management of cystoid macular edema secondary to retinitis pigmentosa via subliminal micropulse yellow laser. Lasers Med Sci. 2021 Mar;36(2):317-323. doi: 10.1007/s10103-020-03031-0. Epub 2020 May 4. PMID 32363437